CLINICAL TRIAL: NCT07221799
Title: A Pilot Study of the Pharmacodynamics and Clinical Effects of Oral Extended Release (OER) Glibenclamide in Multiple Sclerosis Patients With Neuropathic Pain
Brief Title: OER Glibenclamide for Neuropathic Pain in Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00115908
Record Dates: First submitted 2025-10-17; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis; Neuropathic Pain
MeSH Terms: conditions — Multiple Sclerosis; Neuralgia | interventions — Glyburide

STUDY DESIGN:
Intervention Model Description: This is a 2-stage pilot study of the pharmacodynamics and clinical effects of OER glibenclamide in MS patients with neuropathic pain. This pilot study will include 10 subjects. In Stage 1 of the study, which will last 5 days, unblinded subjects will take test-drug twice daily each day and participate in PK determinations. Successful completion of this Stage will establish the ability of a subject to safely tolerate the test-drug. In Stage 2 of the Study, which will last 3 months, blinded subjects who have demonstrated the ability to safely tolerate the test-drug will be asked to evaluate its clinical efficacy specifically with regard to neuropathic pain. By using a 3-block/on-off design with blinding, each subject will serve as their own control during the Stage-2 efficacy part of the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: In stage 2, medication will be either placebo or treatment, blinded in appearance. Investigators will not be aware of placebo/treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral extended release glibenclamide (Experimental): 1. Stage 1, Pharmacokinetics/Pharmacodynamics: This will be a 5 day, unblinded evaluation while participants receive OER-glibenclamide
  2. Stage 2, Safety/Efficacy: This part of the study occurs during weeks 2-13, in 3 successive blocks of 4 weeks each. During this stage, group assignments are randomized, and subjects are blinded as to test-drug vs. placebo. Depending on group assignment, exposure to test-drug may occur early (week-2) or later (week-6). In both groups, exposure to placebo occurs for 4 weeks and exposure to drug occurs for 8 successive weeks.
  Interventions: Drug: glibenclamide
- Placebo (Placebo Comparator): 2. Stage 2, Safety/Efficacy: This part of the study occurs during weeks 2-13, in 3 successive blocks of 4 weeks each. During this stage, group assignments are randomized, and subjects are blinded as to test-drug vs. placebo. Depending on group assignment, exposure to test-drug may occur early (week-2) or later (week-6). In both groups, exposure to placebo occurs for 4 weeks and exposure to drug occurs for 8 successive weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: glibenclamide — oral extended release pill
  Other Names: glyburide
  Arms: oral extended release glibenclamide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is an early phase safety evaluation of the use of oral extended release (OER) glibenclamide, which is otherwise known as glyburide, for use as a treatment for neurologic pain in people with multiple sclerosis. Patients will receive medication to assess safety and tolerability.

DETAILED DESCRIPTION:
This is a 2-stage pilot study of the pharmacodynamics and clinical effects of OER glibenclamide in MS patients with neuropathic pain. This pilot study will include 10 subjects. In Stage 1 of the study, which will last 5 days, unblinded subjects will take test-drug twice daily each day and participate in PK determinations. Successful completion of this Stage will establish the ability of a subject to safely tolerate the test-drug. In Stage 2 of the Study, which will last 3 months, blinded subjects who have demonstrated the ability to safely tolerate the test-drug will be asked to evaluate its clinical efficacy specifically with regard to neuropathic pain. By using a 3-block/on-off design with blinding, each subject will serve as their own control during the Stage-2 efficacy part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Diagnosis of multiple sclerosis per the 2017 Revised McDonald Criteria
3. Score of ≥ 19 on the painDETECT questionnaire

Exclusion Criteria:

1. Severe renal disorder from the patient's history (e.g., dialysis) or eGFR of < 30 ml/min.1.73m2
2. Severe liver disease, or ALT > 3 times upper limit of normal or bilirubin >2 times normal
3. Acute ST elevation myocardial infarction, and/or acute decompensated heart failure, and/or QTc > 520 ms, and/or known history of cardiac arrest (PEA, VT, VF, asystole), and/or admission for an acute coronary syndrome, myocardial infarction, or coronary intervention within the past 3 months
4. T2DM treated with insulin or oral medication
5. Blood glucose < 55 mg/dL at enrollment or immediately prior to administration of study drug or a clinically significant history of hypoglycemia.
6. Known sulfonylurea treatment within 7 days. Sulfonylureas include glyburide/glibenclamide (Diabeta, Glynase); glyburide plus metformin (Glucovance); glimepiride (Amaryl); repaglinide (Prandin); nateglinide (Starlix); glipizide (Glucotrol, GlibeneseR, MinodiabR); gliclazide (DiamicronR); tolbutamide (Orinase, Tolinase); glibornuride (Glutril)
7. Known allergy to sulfa or specific allergy to sulfonylurea drugs
8. Known G6PD enzyme deficiency
9. Pregnancy. Women must be either postmenopausal, permanently sterilized or, if ≤50 years old must have a negative test for pregnancy obtained before enrollment
10. Breast-feeding women who do not agree to stop breastfeeding during Study Drug infusion and for 7 days following the end of Study Drug infusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | over 10 hours
  maximum concentration
Safety | Through week 13
  Full reporting of any adverse events on study drug
Cmin | Over 10 hours
  Minimum concentration
AUC | 10 hours
  Area under curve
tmax | 10 hours
  time to maximum concentration
t 1/2 | 10 hours
  time to 1/2 maximum concentration
blood glucose | 10 hours
  blood glucose during 10 hour pharmacokinetic measurements

SECONDARY OUTCOMES:
Change in PROMIS Neuropathic Pain Scale Score | Through week 13
  The questionnaire uses a standard T-score metric, with a mean of 50 and a standard deviation of 10 for a relevant reference population (often the US general population). Higher scores indicate a greater level of neuropathic pain qualities.
Change in the PROMISE Pain Interference Score | Through week 13
  The PROMIS Pain Interference (PROMIS-PI) scale is a patient-reported outcome measure that assesses how pain affects daily life, including physical, mental, and social activities, as well as sleep and enjoyment. Scores are typically presented on a T-score metric, where 50 is the U.S. general population mean, with higher scores indicating greater pain interference.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Harrison, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No